CLINICAL TRIAL: NCT07143760
Title: Healing Response of Recipient and Donor Sites in Smokers and Non-Smokers Following Free Gingival Grafting: Adjunctive Effects of Topical Hyaluronic Acid on Palatal Healing
Brief Title: Topical Hyaluronic Acid Adjunctive Effects on Healing After Free Gingival Grafting in Smokers and Non-Smokers
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: Ricerfarma S.r.l (Other)
Responsible Party: Principal Investigator, Emine Çifcibaşı, Associate Professor, Istanbul University
Other Study IDs: 2023/18
Record Dates: First submitted 2025-08-06; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Recession, Gingival; Tissue Grafts
Keywords: free gingival graft; hyaluronic acid; smoking; visual analogue scale
MeSH Terms: conditions — Gingival Recession; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Non-smokers who did not use Hyaluronic acid gel: This group consist subjects with Non-smokers who did not use Hyaluronic acid gel
- Non-smokers who used Hyaluronic acid gel: This group consist subjects with Non-smokers who used Hyaluronic acid gel
  Interventions: Device: Gengigel
- Smokers who did not use Hyaluronic acid gel: This group consist subjects with Smokers who did not use Hyaluronic acid gel
- Smokers who used Hyaluronic acid gel: This group consist subjects with Smokers who used Hyaluronic acid gel
  Interventions: Device: Gengigel

INTERVENTIONS:
Device: Gengigel — Free gingival graft (FGG) surgery leaves an open wound at the palatal donor site, which heals by secondary intention and can cause patient discomfort. Various adjunctive materials, such as stents, collagen sponges, platelet-rich fibrin, and hyaluronic acid (HA), have been explored to improve healing. HA is a naturally occurring glycosaminoglycan with hydrating, anti-inflammatory, and pro-regenerative properties that support fibroblast and keratinocyte activity and promote angiogenesis. These qualities make HA a promising adjunct for enhancing wound healing in periodontal surgery. However, few studies have assessed its clinical impact on palatal donor site healing after FGG, and in existing studies HA was applied only once by the operator rather than used consistently by patients. This study evaluates daily, patient-applied HA gel to address this gap and compare outcomes in smokers and non-smokers.
  Groups: Non-smokers who used Hyaluronic acid gel; Smokers who used Hyaluronic acid gel

SUMMARY:
Comparison of the healing of free gingival grafts applied to smokers and non-smokers and evaluation of the effect of hyaluronic acid gel on healing of the donor site.

DETAILED DESCRIPTION:
The oral mucosa consists of three main components: (1) masticatory mucosa, (2) specialized mucosa, and (3) lining mucosa. The masticatory mucosa is a keratinized tissue covering the gingiva and the hard palate. The gingiva itself can be classified into three distinct regions: (1) free gingiva, (2) interdental gingiva, and (3) attached gingiva. The free gingiva is composed of oral epithelium, oral sulcular epithelium, and junctional epithelium. Both the oral epithelium, interdental gingiva, and attached gingiva are keratinized tissues.

Keratinized gingiva can be histologically divided into the following cell layers based on the degree of keratin-producing cell differentiation:

Stratum basale (or stratum germinativum)

Stratum spinosum

Stratum granulosum

Stratum corneum

The absence of keratinized gingiva is classified under mucogingival deformities. These deformities represent deviations from the normal dimensional and morphological relationship between the gingiva and the alveolar mucosa and can often have negative esthetic and functional implications for patients. The lack of keratinized gingiva is addressed separately within mucogingival conditions.

In cases where patients present with a thin gingival biotype, inflammation and gingival recession can further reduce the protective capacity of the tissue, creating clinical scenarios in which mucogingival therapy should be considered. Lang and Löe suggested that an apico-coronal width of keratinized gingiva of less than 2 mm is insufficient to maintain gingival health. Today, the presence of attached gingiva is regarded as crucial for maintaining periodontal health. From a periodontal perspective, keratinized gingiva serves two primary functions:

Providing mechanical resistance against functional forces.

Offering a stable surface for toothbrushing, thus facilitating plaque control.

The 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions concluded that, although a minimum amount of keratinized tissue may not be required to prevent attachment loss when optimal plaque control is achieved, approximately 2 mm of keratinized tissue and 1 mm of attached gingiva around the teeth is considered necessary to maintain periodontal health.

The Free Gingival Graft (FGG) procedure, first described by Björn in 1963, is a surgical technique developed to increase the dimensions of keratinized tissue around teeth and prevent gingival recession. This method remains one of the most commonly employed approaches for augmenting keratinized gingiva. However, over time, transplanted tissue can undergo horizontal and vertical dimensional changes. This makes the long-term volumetric stability of keratinized gingiva after FGG procedures critical. Postoperative graft shrinkage is considered a clinical phenomenon that mainly occurs during the early healing phase.

During FGG surgery, a graft is harvested from the palatal donor site, which is then left to heal by secondary intention. The most frequently observed postoperative complications at the donor site include pain, burning sensation, delayed wound healing, and associated difficulties in eating. Over the years, various hemostatic agents, periodontal dressings, platelet-rich fibrin, and analgesics have been used to reduce these complications and support healing; however, no ideal material has been identified in the literature.

The mechanisms by which smoking affects periodontal status are not fully understood, but numerous potential pathways have been discussed in the literature, including effects on the oral microbiota, gingival tissues, inflammatory and immune responses, and the healing capacity of the periodontium. Although smoking does not directly influence plaque accumulation, it is widely accepted that it can impair various aspects of the innate immune response. In periodontitis, the balance between plaque and immune response may shift toward exaggerated tissue destruction, meaning that even a small amount of plaque can lead to disproportionate breakdown.

Evidence suggests that, in smokers, the function and adhesion of gingival and periodontal ligament fibroblasts may be compromised, collagenolytic activity may increase, and collagen production may decrease. Additionally, the suppression of gingival inflammation, reduction in bleeding on probing, and decreased gingival bleeding seen in smokers are not due to vasoconstriction of the gingival vasculature but rather to reduced angiogenesis within the tissues.

For these reasons, mucogingival problems are more prevalent among smokers, with a clear dose-response relationship. Smoking may also negatively impact both the short- and long-term success of periodontal plastic surgery procedures. As a result, the expected dimensions of keratinized gingiva at the recipient site may not be achieved, and smokers may face a higher risk of postoperative complications.

In a study smoking did not appear to have a noticeable impact on postoperative dimensional changes of FGG, it was shown to reduce postoperative bleeding and delay epithelialization, ultimately slowing donor site wound healing.

Hyaluronic acid (HA) is a high-molecular-weight, non-sulfated polysaccharide of the glycosaminoglycan family, found in various body fluids such as synovial fluid, serum, saliva, and gingival crevicular fluid. HA is present in all periodontal tissues-at higher concentrations in non-mineralized tissues like the gingiva and periodontal ligament and at lower levels in mineralized tissues like cementum and alveolar bone. HA is synthesized by mesenchymal cells such as fibroblasts, chondrocytes, and osteoblasts at the cell membrane.

Because HA is highly biocompatible and non-immunogenic, it has bacteriostatic, fungistatic, anti-inflammatory, anti-edematous, osteoinductive, and pro-angiogenic properties, contributing to wound healing in various tissues. These properties have made HA an attractive adjunct in fields such as orthopedics, ophthalmology, and dermatology for treating a range of conditions.

In dentistry, HA has been applied to accelerate healing in extraction sockets, treat temporomandibular joint osteoarthritis, maintain space in sinus lift procedures without grafting, and relieve pain associated with recurrent aphthous ulcers. In periodontology, HA has been proposed for use either as a monotherapy or as an adjunct to non-surgical and/or surgical periodontal therapy to reduce inflammation and support wound healing.

To the best of our knowledge, there is no study in the literature evaluating the potential effects of HA on VAS scores and healing outcomes specifically in smokers undergoing FGG surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients were eligible for inclusion if they were between 18 and 65 years of age, systemically healthy, and not taking regular medication. Additional criteria included the absence of antibiotic use within the last three months, no pregnancy or lactation, a periodontally healthy status or completion of periodontal therapy, and the presence of insufficient keratinised gingiva in the mandibular anterior region (canine-to-canine) with a clinical indication for FGG in the same area. Smoking and non-smoking status were determined from clinical records and patient self-reports. All smokers included in the study continued smoking throughout the documented postoperative period, and none of the non-smokers had a history of smoking or initiated smoking during the study period.

Exclusion Criteria:

Subjects who do not meet these conditions will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After screening archived patient records from the Istanbul University, Dentistry Faculty, Department of Periodontology archive, a total of 80 patients who had undergone FGG surgery between January 2018 and November 2022 were deemed eligible and included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Healing outcome of the palatal donor site | Baseline, Day 7 , Day 14, 1. Month, 3. Months
  Clinical assessment of epithelialisation using standardised scoring. Assessment of the palatal donor site was undertaken through standardised measurements of graft epithelialisation at predefined intervals using a Williams periodontal probe.

SECONDARY OUTCOMES:
Visual Analogue Scale pain scores | Days 3, 7, 10, and 14 postoperatively
  Patient-reported pain levels measured using a 10-cm visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Dentistry Faculty, Department of Periodontology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yildirim S, Ozener HO, Dogan B, Kuru B. Effect of topically applied hyaluronic acid on pain and palatal epithelial wound healing: An examiner-masked, randomized, controlled clinical trial. J Periodontol. 2018 Jan;89(1):36-45. doi: 10.1902/jop.2017.170105. PMID 28914592
- [Background] Silva CO, Ribeiro Edel P, Sallum AW, Tatakis DN. Free gingival grafts: graft shrinkage and donor-site healing in smokers and non-smokers. J Periodontol. 2010 May;81(5):692-701. doi: 10.1902/jop.2010.090381. PMID 20429648
- [Background] Hatipoglu H, Keceli HG, Guncu GN, Sengun D, Tozum TF. Vertical and horizontal dimensional evaluation of free gingival grafts in the anterior mandible: a case report series. Clin Oral Investig. 2007 Jun;11(2):107-13. doi: 10.1007/s00784-006-0084-x. Epub 2007 Feb 9. PMID 17294229
- [Background] Cifcibasi E, Karabey V, Koyuncuoglu C, Duzagac E, Genceli E, Kasali K, Cintan S. Clinical evaluation of free gingival graft shrinkage in horizontal and vertical dimensions. J Istanb Univ Fac Dent. 2015 Oct 21;49(3):11-16. doi: 10.17096/jiufd.58759. eCollection 2015. PMID 28955540
- [Background] Björn, H. (1963). Free Transplantation of Gingiva Propria. Odontol. Rev.